CLINICAL TRIAL: NCT06103409
Title: Allogenic Mesenchymal Stromal Cells for the Treatment of Burn Wounds.
Brief Title: MSCs for the Treatment of Burn Wounds
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto Venezolano de Investigaciones Cientificas (Other)
Collaborators: Unidad de Terapia Celular - IVIC (Unknown); Hospital Pediátrico Niño Jesús, San Felipe, Yaracuy (Unknown); Hospital Central Dr. Plácido D. Rodriguez Rivero, San Felipe, Yaracuy (Unknown)
Responsible Party: Principal Investigator, Dylana Diaz Solano, Investigator, Instituto Venezolano de Investigaciones Cientificas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVIC-UTC-MSC-Burn
Record Dates: First submitted 2023-10-23; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Burn Wound; Second- or Third-degree Burn
Keywords: Burn wounds, skin regeneration, MSCs
MeSH Terms: conditions — Burns; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogenic MSCs (Experimental): All Patients will receive conservative treatment before transplantation of allogenic MSCs embedded in autologous platelet rich plasma clot.
  Interventions: Biological: Implantation of allogeneic MSCs on burn wounds

INTERVENTIONS:
Biological: Implantation of allogeneic MSCs on burn wounds — Transplantation of allogeneic MSCs in patients with deep- or full-thickness burns. Allogeneic MSCs embedded in autologous platelet rich plasma clot (PRP) are implanted onto the burned areas. The treated areas will be covered with conventional dressings and burned roll. Dressings will be changed after 5 days and then weekly. The total number of MSCs used in each patient varied according to the burn injury. In patients with larger burned areas, its necessary to apply new treatments with MSCs in affected areas, at intervals of at least 1 month. Implantation will be performed in the operating room. Patients will receive first line treatments.
  Other Names: Transplantation of MSCs on burn wounds

SUMMARY:
The goal of this study is to evaluate the capacity of allogenic mesenchymal stromal cells form bone marrow (BM-MSC) or adipose tissue(Ad-MSC) to induce wound healing in patients with burn wounds.

DETAILED DESCRIPTION:
Based on the paracrine and immunomodulatory effects of MSCs, they are considered promising cells for tissue engineering and skin regeneration in burn wounds. This protocol is designed to evaluate the efficacy of transplantation of allogenic BM-MSCs or Ad-MSCs, included in preclotted platelet-rich plasma (PRP), in patients with deep- or full-thickness burns (second- or third-degree / AB B or B degree). All patients will receive concomitant first-line treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 weeks and 85 years old
* Patient with second- or third-degree burn (AB/B or B).
* Thermal burns
* Electrical burns
* Chemical burns
* Informed consent of the patient or caretaker

Exclusion Criteria:

* First degree burn (A or AB)
* Evidence of active infection at the wound site
* Chronic malnutrition
* Systemic inflammatory response syndrome (SIRS) or sepsis
* Moderate or severe respiratory tract or lungs burn injuries
* Autoimmune disease (e.g. multiple sclerosis, lupus erythematosus)
* Severe pulmonary disease, hematologic disease, malignancy, or hypo-immunity.
* Diabetes
* Pregnancy

Ages: 2 Weeks to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Re-epithelialization areas | Up to 6 month
  Re-epithelialization will be determined by clinical evaluations and recorded by digital color photographs
Complete burn wound healing | Up to 12 month
  Time (days) to complete re-epithelialization of burned skin. It will be based on clinical evaluations and digital color photographs

CONTACTS AND LOCATIONS:
Overall Officials: Olga L Wittig, MSc, Principal Investigator — Instituto Venezolano de Investigaciones Cientificas
Locations (1):
- Instituto Venezolano de Investigaciones Cientificas, Caracas, Miranda, Venezuela

REFERENCES:
- [Background] Wittig O, Diaz-Solano D, Chacin T, Rodriguez Y, Ramos G, Acurero G, Leal F, Cardier JE. Healing of deep dermal burns by allogeneic mesenchymal stromal cell transplantation. Int J Dermatol. 2020 Aug;59(8):941-950. doi: 10.1111/ijd.14949. Epub 2020 Jun 5. PMID 32501530
- [Background] Pereira B, Duque K, Ramos-Gonzalez G, Diaz-Solano D, Wittig O, Zamora M, Gledhill T, Cardier JE. Wound healing by transplantation of mesenchymal stromal cells loaded on polyethylene terephthalate scaffold: Implications for skin injury treatment. Injury. 2023 Apr;54(4):1071-1081. doi: 10.1016/j.injury.2023.02.024. Epub 2023 Feb 13. PMID 36801131
- [Background] Ramos-Gonzalez G, Salazar L, Wittig O, Diaz-Solano D, Cardier JE. The effects of mesenchymal stromal cells and platelet-rich plasma treatments on cutaneous wound healing. Arch Dermatol Res. 2023 May;315(4):815-823. doi: 10.1007/s00403-022-02451-y. Epub 2022 Nov 3. PMID 36326886
- [Background] Ramos-Gonzalez G, Wittig O, Diaz-Solano D, Salazar L, Ayala-Grosso C, Cardier JE. Evaluation of epithelial progenitor cells and growth factors in a preclinical model of wound healing induced by mesenchymal stromal cells. Biosci Rep. 2020 Jul 31;40(7):BSR20200461. doi: 10.1042/BSR20200461. PMID 32667622